CLINICAL TRIAL: NCT06323148
Title: Adjuvant Target Therapy Guided by ctDNA-MRD in Patients With EGFR-mutant II-IIIA
Brief Title: Adjuvant Target Therapy Guided by ctDNA-MRD in Patients With EGFR-mutant II-IIIA Non-small Cell Lung Cancer (ECTOP-1022)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-1022
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; EGFR Gene Mutation; Minimal Residual Disease
MeSH Terms: conditions — Lung Neoplasms; Neoplasm, Residual | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ct-DNA-positive patients receiving no adjuvant osimertinib (Placebo Comparator): ct-DNA-positive patients receiving no adjuvant osimertinib
  Interventions: Drug: No adjuvant therapy
- ct-DNA-positive patients receiving adjuvant osimertinib (Experimental): ct-DNA-positive patients receiving adjuvant osimertinib
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Adjuvant osimertinib for three years after radical surgery
  Arms: ct-DNA-positive patients receiving adjuvant osimertinib
Drug: No adjuvant therapy — No adjuvant therapy
  Arms: ct-DNA-positive patients receiving no adjuvant osimertinib

SUMMARY:
This study plans to conduct ctDNA testing on EGFR mutation-positive stage II-IIIA (N1-N2) NSCLC patients after radical surgery (R0 resection). Patients with positive ctDNA testing will receive standard treatment according to clinical guidelines, while patients with negative ctDNA testing will be assessed based on comprehensive clinical and pathological characteristics. After receiving or not receiving standard adjuvant chemotherapy, patients will be randomly assigned in a 1:1 ratio to either the observation follow-up group (experimental group) or the osimertinib adjuvant treatment group (control group). The aim is to explore whether observation follow-up for patients with negative ctDNA after surgery has a prognosis non-inferior to osimertinib treatment, and to investigate the disease-free survival rate of EGFR mutation-positive stage II-IIIA (N1-N2) NSCLC patients with positive ctDNA after surgery receiving osimertinib adjuvant treatment, providing more precise treatment guidance for adjuvant therapy in this specific type of NSCLC patients with EGFR mutation-positive tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years old, both males and females are eligible.
2. Histologically confirmed diagnosis of non-small cell lung cancer.
3. Diagnosis of stage II-IIIA (N1-N2) non-small cell lung cancer based on the 8th edition TNM staging guidelines combined with radiological evaluation.
4. EGFR mutation-positive status confirmed through molecular testing (such as ARMS-PCR or high-throughput sequencing), specifically with mutations 19del or 21L858R.
5. Able to undergo R0 surgical resection.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-1. Expected survival of more than 12 months.
7. Baseline blood routine and biochemical indicators meeting the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   * Lymphocyte count ≥ 0.5 × 10^9/L;
   * Platelet count ≥ 100 × 10^9/L;
   * Hemoglobin ≥ 9 g/dL.
   * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 times ULN.
8. Patients must provide informed consent, either directly or through their legally authorized representatives, after being informed about the study.

Exclusion Criteria:

1. Pathological diagnosis of mixed-type lung cancer (including a history of small cell lung cancer or non-adenocarcinoma).
2. Received anti-tumor therapy before surgery (including radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.).
3. Rx, R1, R2 surgical resection.
4. Received blood transfusion during surgery or within 2 weeks before surgery.
5. Pregnant or lactating female patients.
6. History of other malignant tumors within the past 5 years, except for cases where other malignant tumors have been cured solely through surgery with a disease-free interval of at least 10 years, curable basal cell carcinoma of the skin, and cervical carcinoma in situ.
7. Any unstable systemic diseases (including active infections, uncontrolled hypertension, unstable angina pectoris, congestive heart failure, myocardial infarction within the past year, severe arrhythmias requiring medication, liver, kidney, or metabolic diseases).
8. Evidence of any other diseases, neurological or metabolic functional disorders, physical examination findings, or laboratory findings that would place the subject at high risk of treatment-related complications.
9. Other factors deemed by the investigators to potentially affect the study process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The 3-year Disease-Free Survival (DFS) rate between the observation group and the osimertinib treatment group. | 3 years
  Disease-Free Survival

IPD SHARING:
Plan to Share IPD: Undecided